CLINICAL TRIAL: NCT03307746
Title: A Phase IIa Study of RItuximab and VArlilumab in Relapsed or Refractory B-cell Malignancies
Brief Title: A Combination of Rituximab and Varlilumab Immunotherapy in Patients with B-cell Lymphoma
Acronym: RiVa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University Hospital Plymouth NHS Trust (Other); The Christie NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Celldex Therapeutics (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAN1278
Record Dates: First submitted 2017-08-07; First posted 2017-10-12 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — varlilumab; Rituximab

STUDY DESIGN:
Intervention Model Description: Patient will be randomised into Arm A (20 patients) or Arm B (20 Patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A- Rituximab and Varlilumab (Active Comparator): Patients in ARM A willl receive Cycle1 Day 1: rituximab 375 mg/m2 IV Cycle 1 Day 2: varlilumab 3 mg/kg IV Cycles 2 Day 1: rituximab 375 mg/m2 IV Cycle 3 Day 1: rituximab 375 mg/m2 IV Cycle 3 Day 2: varlilumab 3 mg/kg IV Cycle 4 Day 1: rituximab 375 mg/m2 IV Cycle 5 Day 1: rituximab 375 mg/m2 IV Cycle 5 Day 2: varlilumab 3 mg/kg IV Cycle 6 Day 1: rituximab 375 mg/m2 IV
  Interventions: Drug: Varlilumab
- ARM B - Rituximab and Varlilumab (Active Comparator): Patients in ARM B will receive Cycle 1 Day 1: rituximab 375 mg/m2 IV Cycle 1 Day 8: varlilumab 3 mg/kg IV Cycle 2 Day 1: rituximab 375 mg/m2 IV Cycle 3 Day 1: rituximab 375 mg/m2 IV Cycle 3 Day 2: varlilumab 3 mg/kg IV Cycle 4 Day 1: rituximab 375 mg/m2 IV Cycle 5 Day 1: rituximab 375 mg/m2 IV Cycle 5 Day 2: varlilumab 3 mg/kg IV Cycle 6 Day 1: rituximab 375 mg/m2 IV
  Interventions: Drug: Varlilumab

INTERVENTIONS:
Drug: Varlilumab — Rituximab is a so-called direct-targeting mAb, which binds to the CD20 molecule on the surface of normal and malignant B cells. The mAb then engages immune effectors cells, such as macrophages, through Fc:Fc gamma receptor interaction, leading to tumour cell killing by antibody directed cellular cytotoxicity and/or phagocytosis (ADCC/ADCP).
  Varlilumab (1F5, CDX-1127) is a recombinant and fully human IgG1kappa mAb that binds to human CD27 with high affinity (62). As far as we are aware, it is the only anti-CD27 mAb in clinical development. Once bound, varlilumab blocks CD70 binding to CD27.
  Other Names: Rituximab

SUMMARY:
A total of 40 participants will be recruited, with 20 participants in each of the following subcategories:

A) High grade lymphoma (DLBCL, FL grade 3b, transformed FL) (n=20) B) Low grade lymphoma (e.g. FL grade 1, 2 or 3a, MZL, MCL) (n=20)

The main purpose for having two experimental treatment arms is to provide a comparator for the translational endpoints, i.e. to assess whether the differences observed are due to the addition of varlilumab to rituximab. The only difference between Arm A and Arm B is the delay in administration of varlilumab in cycle 1, which is on Day 2 in Arm A and Day 8 in Arm B. As the post-treatment tissue collection occurs on Day 7/8, prior to administration of varlilumab in Arm B, samples will be obtained from participants that have either been treated with rituximab alone, or both rituximab and varlilumab. To minimise any potential risks to the patient as a result of a repeat biopsy on Day 7/8, a prerequisite for entry to the trial is that the participants must have accessible sites for biopsy. Difference in response rates between Arm A and Arm B are not expected.

DETAILED DESCRIPTION:
A multicentre, randomised, phase IIa study in participants with relapsed or refractory CD20+ B-cell malignancies. The study will be conducted in 2 stages as follows:

Stage 1 - Safety During the safety phase, 6 participants (3 from each Arm and from any subtype) will be treated as detailed in section 6.1. The number of dose limiting toxicities (DLTs) experienced by these participants in each arm after having completed the first cycle will dictate whether the trial will proceed to the second stage.

1. In each arm, if out of these 3 participants 0 experience a DLT, then that arm will proceed to stage 2.
2. In each arm, if out of these 3 participants 1 or 2 experience a DLT, then that arm will be expanded to 3 more participants.

   1. If 1 or 2 out of 6 participants experience a dose limiting toxicity, the arm will proceed to Stage 2.
   2. If 3 or more out of 6 participants experience a DLT, recruitment for that arm will be stopped.
3. If out of these 3 participants, 3 experience a dose limiting toxicity, recruitment for that arm will be stopped.

Initially, the first patient will be entered into the trial. Providing there are no serious or unexplained safety issues during the first 2 weeks, as determined by the Safety Review Committee (SRC), then dosing of subsequent participants will continue as they are identified. Should toxicity findings of concern occur, the SRC may choose to stagger the start of dosing for subsequent participants and/or cohorts.

The objective of Stage 2 is to obtain some further information on the safety of the intervention in a larger sample, information on activity (response rate overall and per lymphoma subtype) and feasibility of administrating rituximab and varlilumab together. During Stage 2, recruitment will continue so (including those in Stage 1), there is a total of 10 participants per arm and per disease category (a total of 20 participants per disease category, 40 participants in the trial in total).

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory CD20+ B-cell lymphoma excluding chronic lymphocytic leukaemia/small lymphocytic lymphoma (CLL/SLL).

   * High grade subgroup: Diffuse large B-cell lymphoma, FL grade 3b, transformed FL
   * Low grade subgroup: All low grade CD20+ B-cell lymphoma subtypes excluding CLL/SLL (e.g. FL grade 1,2 or 3a, MCL, LPL)
2. Disease must be recurrent or treatment refractory, and received at least one line of treatment. Rituximab-refractory participants are eligible for the entry into the study as long as the tumour expresses CD20.
3. At least one measurable lesion by CT scan (defined as >1.5 cm in one axis) that is also easily accessible for biopsy.
4. Histological confirmation of relapse within 12 months of treatment.
5. 16 years of age or older.
6. Haematological and biochemical indices with the ranges shown below:

   * Laboratory Test Value required

     * Haemoglobin (Hb) ≥ 90 g/L (red cell support is permissible)
     * Absolute neutrophil count (ANC) ≥1.0 x 109/L (or ≥0.5 x 109/L if bone marrow involvement) G-CSF support is not permissible at screening.
     * Platelet count ≥75 x 109/L (or ≥30 x 109/L if bone marrow involvement)
     * Serum bilirubin ≤1.5 x upper limit of normal (ULN) unless raised due to Gilbert's syndrome in which case up to 3 x ULN is permissible
     * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x ULN unless raised due to hepatic involvement
     * Calculated creatinine clearance (Cockcroft-Gault formula) ≥30 ml/min (uncorrected value)
7. Ability to understand the purpose and risks of the study and provide written informed consent .
8. Willing and able to participate in all required evaluations and procedures in this study protocol.
9. Participants must be willing to participate in appropriate pregnancy prevention measures:

   * Women of childbearing potential who have a negative serum or urine pregnancy test during screening (within 14 days prior to the start of trial treatment) and agree to use one highly effective form of contraception combined with an effective form of contraception (see below) effective from the first administration of all study drugs, throughout the trial and for 12 months after last dose all study drugs are considered eligible.
   * Male participants with partners of child-bearing potential who agree to take measures not to father children by using one form of highly effective contraception from the first administration of all study drugs, throughout the trial and for 12 months after last dose of all study drugs are considered eligible. Male subjects must also refrain from donating sperm during this period.

   Contraception

   Contraception that is considered highly effective includes oral, injected or implanted progesterone-only hormonal contraception (with inhibition of ovulation); oral, intravaginal, or transdermal combined (oestrogen and progesterone containing) hormonal contraception (with inhibition of ovulation); an intra-uterine device (IUD); an intrauterine hormone releasing system (IUS); bilateral tubal occlusion; vasectomised partner or abstinence.

   Contraceptive methods considered to be effective include progesterone-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action; condom; cap, diaphragm or sponge with spermicidal gel.
   * Men with pregnant or lactating partners must be advised to use barrier method contraception (for example: condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
10. Life expectancy ≥ 12 weeks.
11. ECOG performance status 0-2.

Exclusion Criteria:

1. Known central nervous system involvement by lymphoma, that is not in remission, are excluded from the study.
2. History of other malignancy within the last 2 years except for:

   * Noninvasive malignancies such as adequately treated ductal carcinoma in situ of the breast, non-melanoma skin cancer or lentigo maligna, cervical carcinoma in situ and urothelial papillary noninvasive carcinoma or carcinoma in situ, and
   * Prostate intraepithelial neoplasia without evidence of prostate cancer.
3. Receiving treatment (or within a month of) with chemotherapy, immunotherapy or immunosuppressive agents. This includes any systemic steroids at dose exceeding 10 mg prednisolone (or other steroid equivalent) within 2 weeks prior to first dose of varlilumab.
4. Significant concurrent, uncontrolled medical condition that in the opinion of the Investigator contraindicates participation in this study.
5. Active and documented autoimmune disease (including, but not limited to, inflammatory bowel disease, coeliac disease, haemolytic anaemia, or immune thrombocytopenic purpura) prior to first dose of varlilumab.
6. Active infection requiring systemic therapy.
7. Women who are pregnant or lactating.
8. Serological positivity for Hepatitis B, C, or known HIV infection. As per standard of care the results of hepatitis serology should be known prior to commencement of immunochemotherapy.

   * Positive test results for chronic HBV infection (defined as positive HBsAg serology and positive HBcAb) will not be eligible. Participants with occult or prior HBV infection (defined as negative HBsAg and positive HBcAb) will not be eligible. Participants who have protective titres of hepatitis B surface antibody (HBsAb) after vaccination will be eligible.
   * Positive test results for hepatitis C (HCV antibody serology testing) will not be eligible.
9. Previous recipient of an allogeneic bone marrow transplant at any time.
10. Autologous bone marrow transplant within 100 days of first dosing.
11. Systemic radiation therapy within 4 weeks or prior focal radiotherapy within 2 weeks prior to first dosing.
12. Subjects known or suspected of being unable to comply with the protocol.
13. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1-toxicities, which in the opinion of the Investigator should not exclude the patient.
14. Uncontrolled congestive cardiac failure, cardiac ischaemia or cardiac arrhythmia. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to registration, congestive heart failure (NYHA III-IV).
15. Subjects with a known hypersensitivity to rituximab (≥Grade 3) or murine proteins, or any other excipients used in the formulation of rituximab.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Causality and severity of each adverse event | From date of consent, up to max. 15 months
  Causality of each adverse event and grading of severity according to NCI CTCAE version 4.03
Activity - Lugano response criteria | 4 months
  Response of disease to treatment assessed at the end of treatment via contrast enhanced CT scan and classified according to the Lugano Revised Response Criteria for Malignant Lymphoma

SECONDARY OUTCOMES:
Overall Survival | Time from randomisation until death from any cause up to a max. of 15 months after randomisation
  Survival status will be assessed every 2 months
Progression-Free Survival | Time from randomisation until disease progression or death from any cause up to a max. of 15 months after randomisation
  Length of time that patients are free from disease

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No